CLINICAL TRIAL: NCT05027490
Title: Impact of a Nutritional, Sensory and Culinary Support on the Improvement of the Quality of Life Related to Meals in Patients With Cancer Cancer Patients Treated With Chemotherapy
Brief Title: CAncer, NUtrition and Taste 2
Acronym: CANUT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_0409
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Gynecologic Cancer; Bronchial Cancer; Breast, Gynecological or Bronchial Cancer Treated With Intravenous Chemotherapy
Keywords: cancer; nutrition; food perceptions alterations
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Bronchogenic; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients receiving CANUT support (guide + dietary interviews) (Experimental): Patients included in this arm will have following interventions :
  * CANUT support : patients will receive the CANUT guide (food guide) to help them deal with eating disorders encountered during their chemotherapy treatment ; the CANUT support includes calls from a dietician between chemotherapy cycles for support and advice.
  * anthropometric measures
  * Prehension strength measurement
  * food quality of life questionnaire (Qualité de Vie Alimentaire QVA)
  * Quality of Life Questionnaire Core 30 (QLQ C30)
  * Scratch & Snif Test
  * Taste Strip Test
  * Nutrition interview
  * 24 H feed back questionnaire
  * condiment questionnaire
  * tobacco questionnaire
  Interventions: Other: CANUT support; Other: Anthropometric measures; Other: Prehension strength measurement; Behavioral: QVA Questionnaire; Behavioral: QLQ C30 Questionnaire; Behavioral: Scratch & Snif Test; Behavioral: Taste Strip Test; Behavioral: 24 H feed back questionnaire; Behavioral: Condiment questionnaire; Behavioral: Tobacco questionnaire; Other: Nutrition interview
- patients not receiving canut support (guide + dietary interviews) (Active Comparator): Patients included in this arm will have following interventions :
  * anthropometric measures
  * Prehension strength measurement
  * food quality of life questionnaire (Qualité de Vie Alimentaire QVA)
  * Quality of Life Questionnaire Core 30 (QLQ C30)
  * Scratch & Snif Test
  * Taste Strip Test
  * Nutrition interview
  * 24 H feed back questionnaire
  * condiment questionnaire
  * tobacco questionnaire
  Interventions: Other: Anthropometric measures; Other: Prehension strength measurement; Behavioral: QVA Questionnaire; Behavioral: QLQ C30 Questionnaire; Behavioral: Scratch & Snif Test; Behavioral: Taste Strip Test; Behavioral: 24 H feed back questionnaire; Behavioral: Condiment questionnaire; Behavioral: Tobacco questionnaire; Other: Nutrition interview

INTERVENTIONS:
Other: CANUT support — CANUT support includes delivery of the CANUT guide (food guide developed by Paul Bocuse Institute from previous results) ; it will be given to patient with explanations about the use of the guide. This also includes 2 calls from a dietician, performed between the 1st and the 3rd chemotherapy cycle to help patient personally with their food side effects.
  Arms: patients receiving CANUT support (guide + dietary interviews)
Other: Anthropometric measures — These measures include weight, waist size, hip size and brachial circumference
Other: Prehension strength measurement — Prehension strength will be assessed thanks to a hand grip device, that makes it possible to measure strength of all fingers, hands, wrists and forearms muscles
Behavioral: QVA Questionnaire — Food quality of life questionnaire
Behavioral: QLQ C30 Questionnaire — Quality of Life questionnaire Core 30
Behavioral: Scratch & Snif Test — The Scratch & Snif Test is used to assess olfactory capacities : patient has to scratch a box on a card, smell it and recognize the scent amongst a list of propositions
Behavioral: Taste Strip Test — The Taste Strip Test is used to assess taste capacities : strips impregnated with different concentrations of the 5 basic taste qualities (sweet, sour, acid, bitter, umami) are successively placed on patient's tongue ; patient has to identify the taste bit by bit.
Behavioral: 24 H feed back questionnaire — This questionnaire describes patient's food and drink intakes during the last 24 ours
Behavioral: Condiment questionnaire — This questionnaire used to assess condiments consumption
Behavioral: Tobacco questionnaire — This questionnaire used to assess tobacco consumption
Other: Nutrition interview — This interview will be conducted by a dietician

SUMMARY:
Although it has been established that the perception of food and eating and cooking habits change during cancer and its treatment, quality of life related to meals, which is an indicator of the psychobiological and physiological well-being of patients in their relationship to food, has been little studied in the pathological context, and particularly in patients undergoing chemotherapy.

Beyond its biological role, food plays a significant psychobiological and social role, as shown by a series of qualitative studies based on interviews with patients. Following a cancer diagnosis, loss of appetite, difficulty in sharing a meal with the family, and reduced pleasure in eating disrupt the patient's relationship with his or her food.

Thus, side effects such as fatigue, nausea and vomiting, and alterations in taste and smell induced by chemotherapy will affect patients' eating behavior, increasing the risk of deteriorating their quality of life with food. As these side effects are less known and therefore less expected by patients, they often lack the information and tools necessary to understand them.

The present study proposes a support for cancer patients treated by chemotherapy in order to improve their quality of life related to meals, and thus keep the pleasure of eating and reduce the risks of malnutrition. This support will consist of a guide provided to patients, in which they will have information on the functioning of the sensory systems involved in the eating experience, advice and culinary tips to adapt foods to their sensory disorders, and recipes that can be adapted in mild (for patients with hypersensitivity to tastes/smells), accentuated (for patients with hypersensitivity to tastes/smells) and enriched (for patients at risk of denutrition) versions. In addition, their sensory abilities will be assessed at the beginning of the study by psychophysical tests, then between each chemotherapy via a telephone interview (self-reported sensory abilities), and they will benefit from orientation according to the test results.

This work will be a first action to improve the quality of life related to the meal by information, follow-up, and adaptation of the meals to the sensory performances of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Major patient with one of the following 3 types of cancer:

  * Stage 4 lung cancer (TNM 7 or 8). The indication for immunotherapy in addition to first line chemotherapy will not be a criterion for non-inclusion patients
  * histologically or cytologically proven localized breast cancer cytologically proven
  * Gynecological cancer (ovarian cancer or uterine cancer) stage III-IV without functional digestive signs related to the tumor disease
* Patient with a body mass index (BMI) between 18 Kg/m² and 35 Kg/m².
* Patient for whom the indication for treatment with a first line of intravenous chemotherapy (+/- targeted therapy) has been accepted by multidisciplinary meeting.
* Patient naive to previous chemotherapy.
* Life expectancy > 3 months.
* Patient with written informed consent
* Patient affiliated to a French social security system.

Exclusion Criteria:

* Patient under 18 years
* Patient who had another malignancy within the last 3 years years, with the exception of carcinoma in situ of the cervix or cervical carcinoma in situ or adequately treated squamous cell carcinoma of the skin adequately treated, or basal cell skin cancer.This cancer must be adequately controlled.
* Patients with symptomatic brain and/or meningeal metastases.
* Patients with symptomatic mucositis.
* Patients suffering or having suffered from an ear, nose and throat disease or oeso-gastro intestinal pathology interfering with the food intake.
* Patients suffering from digestive disorders such as nausea prior to any cancer treatment.
* Indication of concomitant radiotherapy or immunotherapy treatment alone.
* Patients with a known food allergy or intolerance
* Patient with diagnosed partial or total ageusia.
* Patient with diagnosed partial or total anosmia.
* Patient having used artificial feeding in the 2 months prior to inclusion.
* Patient who has lost more than 10% of baseline weight in the 2 months prior to inclusion.
* Patient unable to be regularly followed for any reason (geographical, family, social, psychological,...).
* Patient deprived of liberty or placed under guardianship or legal protection.
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
QVA questionnaire score difference between the 2 arms | At the end of study follow-up, up to 12 weeks
  The main endpoint of CANUT-2 is the comparison of the overall score of the food quality of life questionnaire (Qualité de Vie Alimentaire QVA) between patients who received CANUT support and those who did not receive the CANUT support. The comparison is performed at the time of V2 i.e. after 4 cycles of chemotherapy treatment, corresponding with the end of study follow-up.

SECONDARY OUTCOMES:
QVA questionnaire score | At the end of study follow-up, up to 12 weeks
  Food questionnaire score QVA will be compared for each subsection between the 2 groups and between V1 (inclusion) and V2 (after 4 cycles of chemotherapy), according to the type of cancer.
QLQ-C30 score | At the end of study follow-up, up to 12 weeks
  Quality of life questionnaire score QLQ-C30 will be compared between the 2 arms and between V1 and V2, according to the type of cancer
Weight | At the end of study follow-up, up to 12 weeks
  Anthropometric parameters (weight, waist size, hip size and brachial circumference) associated with 24 H feedback questionnaire score and prehension strength, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer.
waist size | At the end of study follow-up, up to 12 weeks
  Anthropometric parameters (weight, waist size, hip size and brachial circumference) associated with 24 H feedback questionnaire score and prehension strength, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer.
hip size | At the end of study follow-up, up to 12 weeks
  Anthropometric parameters (weight, waist size, hip size and brachial circumference) associated with 24 H feedback questionnaire score and prehension strength, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer.
brachial circumference | At the end of study follow-up, up to 12 weeks
  Anthropometric parameters (weight, waist size, hip size and brachial circumference) associated with 24 H feedback questionnaire score and prehension strength, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer.
Prehension strength | At the end of study follow-up, up to 12 weeks
  This parameter, associated with anthropometric parameters and 24 H feedback questionnaire score, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer
24 H feedback questionnaire score | At the end of study follow-up, up to 12 weeks
  This parameter, associated with anthropometric parameters and prehension strength, will make it possible to assess evolution of nutritional status between the 2 arms and between V1 and V2, according to the type of cancer
Olfactory capacities | At the end of study follow-up, up to 12 weeks
  Olfactory capacities will be assessed thanks to the Scratch & Snif Test
Taste capacities | At the end of study follow-up, up to 12 weeks
  Taste capacities will be assessed thanks to the Taste Strip Test
Trigeminal sensitivity | At the end of study follow-up, up to 12 weeks
  Trigeminal sensitivity will be assessed thanks to a trigeminal sensitivity test
Use of CANUT guide | At the end of study follow-up, up to 12 weeks
  Changes in the frequency of use of the CANUT guide
Patient typology | At the end of study follow-up, up to 12 weeks
  Determining patient typology according to CITAS (Chemotherapy-induced Taste Alteration Scale) scale
Patient satisfaction | At the end of study follow-up, up to 12 weeks
  Determining patient satisfaction using a satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Hôpital Louis Pradel, Service gynécologie, Bron
  - Hôpital Louis Pradel, Service pneumologie, Bron
  - Infirmerie Protestante, Caluire-et-Cuire
  - Hôpital de la Croix Rousse, service pneumologie, Lyon
  - Centre Léon Bérard, service gynécologie, Lyon
  - Centre Léon Bérard, service pneumologie, Lyon
  - Centre hospitalo-universitaire de Lyon Sud, service Oncologie médicale, Pierre-Bénite
  - Centre hospitalo-universitaire de Lyon Sud, service pneumologie, Pierre-Bénite
  - CHU St Etienne,, Saint-Etienne
  - CH de Valence, Valence